CLINICAL TRIAL: NCT02333396
Title: Improving Communication in the Pediatric Intensive Care Unit for Patients Facing Life-Changing Decisions: The Navigate Study
Brief Title: Improving Communication in the PICU: The Navigate Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Kelly Michelson, Kelly Michelson, MD, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: The Navigate Study
Record Dates: First submitted 2015-01-02; First posted 2015-01-07 (Estimated); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Communication
Keywords: Navigator; Intervention Study; Randomized Controlled Trial; Pediatric Intensive Care Unit; Decision Making
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PICU Supports (Experimental): Participants will receive the PICU Supports intervention.
  Interventions: Other: PICU Supports
- Educational Brochure (Active Comparator): Participants will receive an educational brochure about the pediatric intensive care unit.
  Interventions: Other: Educational Brochure

INTERVENTIONS:
Other: PICU Supports — The PICU Supports intervention includes navigator activities and ancillary tools. The Navigator activities include: initial visits with the healthcare team members (HTMs) and parents; weekday visits with the parents and feedback to the HTMs as needed; coordination of weekly family meetings between the parents and HTMs; and support during transitions out of the unit. The ancillary tools include: a PICU handbook; a place for parents to keep track of events and their goals; a provider sheet to inform PICU HTMs about important parental issues, concerns or goals; a bedside communication log so parents know which non-PICU HTMs have visited; an end-of-life checklist; a bereavement packet for those whose child dies; and informational resources.
  Arms: PICU Supports
Other: Educational Brochure — Parents will receive a short educational brochure with information about the pediatric intensive care unit.
  Arms: Educational Brochure

SUMMARY:
The project seeks to study the use of an navigator-based intervention called "PICU Supports." The study will test the impact of PICU Supports during and after PICU discharge on parent outcomes (satisfaction with decision making, decision regret, anxiety, depression, post-traumatic stress, health-related quality of life, and complicated bereavement) and on parent and healthcare team member assessments of communication and team collaboration.

DETAILED DESCRIPTION:
Parents of children admitted to the PICU often face challenging decisions. Research demonstrates deficiencies in communication in the PICU which could impact decision making. This study team has developed a navigator-based intervention call PICU Supports. PICU Supports aims to provide the following types of support to parents of patients in the PICU: emotional; communication (between healthcare team members and parents/families as well as among healthcare team members ); decision making; transitions out of the PICU (i.e. discharge transitions to a non-PICU hospital bed, a long term care facility, or home); and information. Support is accomplished by navigator engagement with parents and healthcare team members and the guided use of navigator supported ancillary tools provided to parents and healthcare team members as needed. During the patient's PICU stay, the navigator activities and use of ancillary tools is directed by the family's needs. Thus PICU Supports uses a predefined framework of activities and tools to provide individualized support directed by the needs of the parent and the patient situation. This research will test PICU Supports in the clinical setting. This will be accomplished by conducting a pilot study of PICU Supports at Ann & Robert H. Lurie Children's Hospital of Chicago (Lurie Children's Hospital), followed by a randomized controlled trial (RCT) comparing the intervention, PICU Supports, to a control, parental receipt of an educational brochure. The RCT will be conducted at Lurie Children's Hospital and at University of Chicago Medicine Comer Children's Hospital (Comer Children's Hospital).

ELIGIBILITY:
Inclusion Criteria:

Case Patients

* patients < 18 years of age admitted to the PICU
* parents are English or Spanish-speakers and who:
* are likely to require PICU care for at least 24 hours (as determined by the PICU attending physician) or
* have a Pediatric Index of Mortality 2 (PIM2) score ≥ 4% (a PIM2 score predicts risk of mortality based on clinical data collected at the time of admission to the PICU)

Case patients will be included in the study if one of his/her parents agrees to participate in the study and signs a written consent form.

Parents of case patients

* Parent of an eligible case patient.
* PICU attending gives permission to approach the parent about the study.
* Parent is an English or Spanish speaker.
* Parent provides written consent for participation.

Healthcare Team Members for the pre-post assessment of team communication and focus group:

-This group will include as many clinicians in the following groups as possible (identified by the site principal investigator): PICU physicians (attendings and fellows); PICU bedside nurses; PICU Advance Practice Nurses (APNs); hospitalists; subspecialty physicians who consult on PICU patients; subspecialty APNs who consult on PICU patients; PICU respiratory therapist; PICU physical/occupational/speech therapists; and social workers (SWs), chaplains, and case managers who follow PICU patients.

Healthcare team members for the written feedback/assessment of the intervention:

-HTMs caring for the case patient at the time of PICU discharge: (PICU attending; PICU fellow; social worker (if involved); chaplain (if involved); bedside nurse; PICU resident, APN or hospitalist; and one to two subspecialty attendings)

Exclusion Criteria:

Exclusion criteria for parents of case patients:

* PICU attending does not give permission to approach the parent about the study.
* Parent is not an English or Spanish speaker.
* Parent does not provide written consent to participate.
* The case patient does not provide assent (if able to provide assent).

Exclusion criteria for Healthcare Team members:

-Healthcare team member that does not regularly care for patients in the PICU.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2015-04-06 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly N Michelson, MD, Principal Investigator — Ann & Robert H. Lurie Childrens Hospital of Chicago
Locations (2):
- United States (2):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The University of Chicago Medicine Comer Children's Hospital, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ashworth RC, Malone JR, Franklin D, Sorce LR, Clayman ML, Frader J, White DB, Michelson KN. Associations of Patient and Parent Characteristics With Parental Decision Regret in the PICU: A Secondary Analysis of the 2015-2017 Navigate Randomized Comparative Trial. Pediatr Crit Care Med. 2024 Sep 1;25(9):795-803. doi: 10.1097/PCC.0000000000003534. Epub 2024 May 10. PMID 38727516
- [Derived] Tager JB, Hinojosa JT, LiaBraaten BM, Balistreri KA, Aniciete D, Charleston E, Frader JE, White DB, Clayman ML, Sorce LR, Davies WH, Rothschild CB, Michelson KN; Navigate Study Investigators. Challenges of Families of Patients Hospitalized in the PICU: A Preplanned Secondary Analysis From the Navigate Dataset. Pediatr Crit Care Med. 2024 Feb 1;25(2):128-138. doi: 10.1097/PCC.0000000000003385. Epub 2023 Oct 27. PMID 37889100

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PICU Supports | Educational Brochure
Started | 224 | 218
Completed | 124 | 117
Not Completed | 100 | 101

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PICU Supports | Educational Brochure | Total
Number analyzed (Participants) | 124 | 117 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (7.6) | 36.4 (8.0) | 35.5 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 3 missing from PICU Supports 4 missing from Informational Brochure
  Participants
    number analyzed (Participants) | 121 | 113 | 234
    Female | 102 | 89 | 191
    Male | 19 | 24 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 12 | 45
  Not Hispanic or Latino | 84 | 98 | 182
  Unknown or Not Reported | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 3 | 9 | 12
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Black or African American | 14 | 25 | 39
  Race: White | 75 | 73 | 148
  Race: More than one race | 0 | 0 | 0
  Race: Unknown or Not Reported | 32 | 10 | 42

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction With Decision Making (Percentage of "Excellent" Scores in the Decision Making Domain of the Pediatric Family Satisfaction in the Intensive Care Unit (pFS-ICU) Questionnaire)
Description: Percentage of "excellent" scores in the decision making domain of the Pediatric Family Satisfaction in the Intensive Care Unit (pFS-ICU) questionnaire; minimum=0, maximum=100, higher score is better outcome
Time Frame: 3-5 weeks following PICU discharge
Measure: Mean (Standard Error); unit: Percentage of "excellent" scores
Arm/Group | PICU Supports | Educational Brochure
Number analyzed (Participants) | 124 | 117
Percentage of "excellent" scores | 60.35 (33.35) | 56.09 (35.23)
Statistical Analysis 1: Comparison: PICU Supports vs Educational Brochure; Test type: Superiority; p = 0.44, Mixed Models Analysis; Beta Estimate = 3.57, 95% CI 2-sided [-5.77 to 12.9], Standard Error of Mean 4.53

2. Secondary Outcome: Pediatric Family Decision Making Satisfaction in the Intensive Care Unit (pFS-ICU)
Description: Measures satisfaction of family who have a child admitted to the Pediatric intensive care unit; Pediatric Family Satisfaction in the Intensive Care Unit (pFS-ICU) questionnaire mean score, range 0-100, higher score is the better outcome
Time Frame: 3-5 weeks following PICU discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PICU Supports | Educational Brochure
Number analyzed (Participants) | 124 | 117
score on a scale | 86.63 (13.28) | 82.8 (17.6)
Statistical Analysis 1: Comparison: PICU Supports vs Educational Brochure; Test type: Superiority; p = 0.09, Mixed Models Analysis; Beta Estimate = 3.62, 95% CI 2-sided [-0.61 to 7.84], Standard Error of Mean 2.05

3. Secondary Outcome: Parental Satisfaction in the PICU (Score on the Pediatric Family Satisfaction in the Intensive Care Unit (pFS-ICU) Questionnaire)
Description: Subscale: Satisfaction with Care Score on the Pediatric Family Satisfaction in the Intensive Care Unit (pFS-ICU) questionnaire; minimum=0, maximum=100, higher score is better outcome
Time Frame: 3-5 weeks after PICU Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PICU Supports | Educational Brochure
Number analyzed (Participants) | 124 | 117
score on a scale | 87.22 (13.43) | 82.94 (17.59)
Statistical Analysis 1: Comparison: PICU Supports vs Educational Brochure; Test type: Superiority; p = 0.05, Mixed Models Analysis; Beta Estimate = 4.13, 95% CI 2-sided [-0.09 to 8.36], Standard Error of Mean 2.05

4. Secondary Outcome: Parental Satisfaction in the PICU (Score on the Pediatric Family Satisfaction in the Intensive Care Unit (pFS-ICU) Questionnaire)
Description: Subscale: Satisfaction with Decision Making Score on the Pediatric Family Satisfaction in the Intensive Care Unit (pFS-ICU) questionnaire; minimum=0, maximum=100, higher score is better outcome
Time Frame: 3-5 weeks after PICU Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PICU Supports | Educational Brochure
Number analyzed (Participants) | 124 | 117
score on a scale | 85.86 (14.94) | 82.59 (19.10)
Statistical Analysis 1: Comparison: PICU Supports vs Educational Brochure; Test type: Superiority; p = 0.19, Mixed Models Analysis; Beta Estimare = 3.02, 95% CI 2-sided [-1.63 to 7.67], Standard Error of Mean 2.26

5. Secondary Outcome: Parental Decision Regret (Decision Regret Scale)
Description: Score on the Decision Regret Scale, a 5-item Likert-scale measure of decision regret; minimum=0, maximum=100; higher score indicates more decision regret
Time Frame: 3-5 weeks after PICU discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PICU Supports | Educational Brochure
Number analyzed (Participants) | 119 | 114
score on a scale | 12.61 (19.89) | 12.87 (16.09)
Statistical Analysis 1: Comparison: PICU Supports vs Educational Brochure; Test type: Superiority; p = 0.93, Mixed Models Analysis; Beta Estimate = -0.22, 95% CI 2-sided [-5.33 to 4.88], Standard Error of Mean 2.47

6. Secondary Outcome: Parental Anxiety (Anxiety SF8a)
Description: Score on the Anxiety Short Form8a, a 8-item Likert-scale measure of anxiety, the higher the score, the worst the anxiety, T-score range of 37.1 - 83.1.
  A T score of 50 is the average fro the US general population. The SD is 10 with a T-score of 60 being 10 worse than the average and a T-score of 40 being 10 better than the average.
Time Frame: 3-5 weeks after PICU discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PICU Supports | Educational Brochure
Number analyzed (Participants) | 123 | 117
score on a scale | 49.32 (9.78) | 49.68 (10.26)
Statistical Analysis 1: Comparison: PICU Supports vs Educational Brochure; Test type: Superiority; p = 0.79, Mixed Models Analysis; Beta Estimate = -0.35, 95% CI 2-sided [-3.02 to 2.31], Standard Error of Mean 1.29

7. Secondary Outcome: Parental Depression (Depression SF8a)
Description: Score on the Depression; Depression Short Form 8a, a 8-item Likert-scale measure of depression; the higher the score, the worst the depression, T-score range of 38.2 - 81.3.
  A T score of 50 is the average fro the US general population. The SD is 10 with a T-score of 60 being 10 worse than the average and a T-score of 40 being 10 better than the average.
Time Frame: 3-5 weeks after PICU discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PICU Supports | Educational Brochure
Number analyzed (Participants) | 123 | 116
score on a scale | 47.71 (8.33) | 47.23 (9.18)

8. Secondary Outcome: Parental Impact of Event/Post-Traumatic Distress (Impact of Event Scale-revised)
Description: A measure of post-traumatic distress; Score on the Impact of Event Scale-revised, a 22-item Likert-scale measure of post-traumatic distress; scale range from 0 - 88; higher numbers mean higher trauma or distress; units on a scale
Time Frame: 3-5 weeks after PICU discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PICU Supports | Educational Brochure
Number analyzed (Participants) | 123 | 116
score on a scale | 14.02 (16.81) | 12.93 (14.32)

9. Secondary Outcome: Parental Health-related Quality of Life (Global Health Scale) Physical
Description: Measure of global physical health; Physical - Score on the Global Health scale, a 10 item Likert-scale measure of overall health-related quality of life; the higher the score the worse global health, t-score range of 16.2 - 67.7.
  A T score of 50 is the average fro the US general population. The SD is 10 with a T-score of 60 being 10 worse than the average and a T-score of 40 being 10 better than the average.
Time Frame: 3-5 weeks after PICU discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PICU Supports | Educational Brochure
Number analyzed (Participants) | 116 | 110
score on a scale | 48.42 (7.50) | 48.9 (7.76)
Statistical Analysis 1: Comparison: PICU Supports vs Educational Brochure; Test type: Superiority; p = 0.64, Mixed Models Analysis; Beta Estimate = 0.49, 95% CI 2-sided [-2.62 to 1.64], Standard Error of Mean 1.03

10. Secondary Outcome: Parental Health-related Quality of Life (Global Health Scale) Mental
Description: Measure of Global Mental Health; Mental - Score on the Global Health scale, a 10 item Likert-scale measure of overall health-related quality of life; high scores indicate worse mental health; T-score range 21.1 - 67.6.
  A T score of 50 is the average fro the US general population. The SD is 10 with a T-score of 60 being 10 worse than the average and a T-score of 40 being 10 better than the average.
Time Frame: 3-5 weeks after PICU discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PICU Supports | Educational Brochure
Number analyzed (Participants) | 116 | 110
score on a scale | 50.02 (8.01) | 50.92 (7.37)
Statistical Analysis 1: Comparison: PICU Supports vs Educational Brochure; Test type: Superiority; p = 0.39, Mixed Models Analysis; Beta Estimate = -0.90, 95% CI 2-sided [-3.02 to 1.22], Standard Error of Mean 1.03

11. Secondary Outcome: Parental Complicated Bereavement (Grief Scale)
Description: Measure of complicated grief in parents after their child's death; Score on the Index of complicated Grief Scale, a 19-item Likert-scale measure of complicated grief; minimum 0, maximum 74; higher numbers mean more complicate grief
Time Frame: 3-5 weeks after PICU discharge
Population: Data from only 4 participants are analyzed because only 4 people whose children died responded to surveys. 3 participants were in the PICU Support arm and 1 in the Educational Brochure Arm. These data are not shown in the Participant Flow Module because of the small numbers.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | PICU Supports | Educational Brochure
Number analyzed (Participants) | 3 | 1
score on a scale | 19 [19 to 19] | 19 [19 to 19]

12. Secondary Outcome: Parent Report of Healthcare Team Satisfaction (Collaboration and Satisfaction About Care Decisions Scale)
Description: Measure of Satisfaction with Healthcare team collaboaration Subscale Collaboration Satisfaction Score of the Collaboration and Satisfaction about Care Decisions scale, 2 items on a 9-item Likert-scale measure of healthcare team communication satisfaction in ICUs, Score range from 2 - 14 with higher numbers meaning more satisfaction
Time Frame: 3-5 weeks after PICU Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PICU Supports | Educational Brochure
Number analyzed (Participants) | 123 | 116
score on a scale | 12.81 (2.01) | 12.09 (2.61)
Statistical Analysis 1: Comparison: PICU Supports vs Educational Brochure; Test type: Superiority; p = 0.13, Mixed Models Analysis; Beta Estiamte = 1.72, 95% CI 2-sided [-0.55 to 3.98], Standard Error of Mean 1.10

13. Secondary Outcome: Parent Report of Healthcare Team Collaboration (Collaboration and Satisfaction About Care Decisions Scale)
Description: Subscale Collaboration Score of the Collaboration and Satisfaction about Care Decisions scale, 7 items on a a 9-item Likert-scale measure of healthcare team communication in ICUs, scale range from 7 - 49. Higher numbers more collaboration.
Time Frame: 3-5 weeks after PICU Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PICU Supports | Educational Brochure
Number analyzed (Participants) | 123 | 116
score on a scale | 44 (6.71) | 42 (9.28)
Statistical Analysis 1: Comparison: PICU Supports vs Educational Brochure; Test type: Superiority; p = 0.13, Mixed Models Analysis; Beta Estimate = 1.72, 95% CI 2-sided [-0.55 to 3.98], Standard Error of Mean 1.10

14. Secondary Outcome: Parental Report of Acceptability and Perceived Effectiveness of PICU Supports (Likert-scale)
Description: Likert-scale items measuring perceived effectiveness and acceptability of the PICU Supports intervention.
  One likert scale item based on previous work. White DB, Cua SM, Walk R, et al. Nurse-led intervention to improve surrogate decision making for patients with advanced critical illness. Am J Crit Care. Nov 2012;21(6):396-409.
  How well did the PICU Supports help with communication in the PICU? scale "Not at all helpful" "Not very helpful" "Somewhat helpful" "Extremely Helpful" "Unable to assess" Scored based on percentage of participants who responded "Somewhat Helpful" or Extremely Helpful"
Time Frame: 3-5 weeks after PICU Discharge
Population: 91.1% (113/124) reported PICU Supports as "extremely" or "somewhat" helpful.
Measure: Count of Participants; unit: Participants
Arm/Group | PICU Supports
Number analyzed (Participants) | 124
Participants | 113

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | PICU Supports | Educational Brochure
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/117
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/117
Other Adverse Events (participants affected / at risk) | 0/124 | 0/117

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-07-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT02333396/Prot_SAP_ICF_000.pdf